CLINICAL TRIAL: NCT00919854
Title: A Phase II, Open Label Trial, to Evaluate Pharmacokinetics, Safety, Tolerability and Antiviral Activity of DRV in Combination With Low-Dose Ritonavir (DRV/Rtv) in Treatment-Experienced HIV-1 Infected Children From 3 Years to Below 6 Years of Age
Brief Title: A Safety Study to Evaluate the Antiviral Activity of Darunavir in Combination With Ritonavir in HIV 1 Infected Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Collaborators: Tibotec Pharmaceutical Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR012553; TMC114-TiDP29-C228 (Other: Tibotec Pharmaceuticals, Ireland)
Record Dates: First submitted 2009-06-11; First posted 2009-06-12 (Estimated); Results first posted 2013-06-24 (Estimated); Last update posted 2014-04-23 (Estimated); Status verified 2014-04

CONDITIONS: Human Immunodeficiency Virus 1
Keywords: Human immunodeficiency virus 1; HIV-1; Darunavir; Ritonavir; Norvir
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Darunavir; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Darunavir (DRV)+Ritonavir (rtv) (Experimental): Before dose adjustment, oral darunavir suspension (100 mg/mL): 20 mg per kg body weight twice daily for children weighing between 10 and <20 kg. After dose adjustment, 25 mg per kg body weight twice daily if weight less than 15 kg, and fixed dose of 375 mg twice daily if weight more than or equal to 15 kg. Before dose adjustment, oral ritonavir solution (80 mg/mL): 3 mg per kg body weight twice daily and after dose adjustment fixed dose of 50 mg twice daily if weight more than or equal to 15 kg.
  Interventions: Drug: Darunavir; Drug: Ritonavir

INTERVENTIONS:
Drug: Darunavir — Darunavir oral suspension (100 mg/mL) will be administered as 20 mg per kg body weight twice daily for children weighing between 10 and <20 kg before dose adjustment. Darunavir oral suspension will be administered 25 mg per kg body weight twice daily if weight less than 15 kg, and fixed dose of 375 mg darunavir tablets twice daily if weight more than or equal to 15 kg after dose adjustment.
Drug: Ritonavir — Ritonavir oral solution (80 mg/mL) will be administered as 3 mg per kg body weight twice daily before dose adjustment and after dose adjustment fixed dose of 50 mg twice daily if weight more than or equal to 15 kg.

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics (what the body does to the medication), safety and antiviral activity to support dose recommendations by body weight of darunavir with low-dose ritonavir (DRV/rtv), in combination with other antiretroviral drugs (ARVs), in treatment-experienced Human immunodeficiency virus 1 (HIV 1) infected children.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), study to evaluate the pharmacokinetics, safety and antiviral activity. Approximately 24 HIV-1 infected children will be enrolled in this study. The study consists of a 4-week screening period, a 48-week treatment period, and a 4-week follow-up period. Participants will receive DRV/rtv according to their body weight. Safety evaluations will include assessment of adverse events, laboratory tests, physical Examination, neurologic examination, vital signs, and electrocardiogram. The total duration of the study will be 56 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a documented HIV 1 infection (by any of the local standard diagnostic methods, such as HIV PCR-DNA, ELISA or western blot (WB) test for HIV antibodies, etc.)
* Body weight from 10 kg to less than 20 kg at screening
* Participants currently on stable ART (anti retroviral therapy) for at least 12 weeks, who need to change their ARV regimen because it is currently failing, with a viral load of greater than 1000 copies/mL
* Screening genotype resistance test results showing less than 3 DRV resistance-associated mutations
* Parents or legal representative willing and able to give consent

Exclusion Criteria:

* Participants with presence of any currently active conditions included in the listing of WHO ( World Health Organisation) Clinical Stage 4 and participants with presence of a non-HIV encephalopathy
* Administration of any ARV (antiretroviral) or non-ARV investigational medication or investigational vaccine within 30 days prior to screening, except for those medications where dose recommendations for children are available
* Life expectancy less than 6 months, according to the judgment of the investigator
* Co-enrollment in other clinical and/or cohort trials without written permission of the Sponsor
* Participants with any active clinically significant disease (eg, tuberculosis [TB], cardiac dysfunction, pancreatitis, acute viral infections) or findings during screening of medical history or physical examination that, in the investigator's opinion, would compromise the subject's safety or outcome of the study

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2009-09; Primary Completion 2010-08 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals, Ireland Clinical Trial, Study Director — Tibotec Pharmaceuticals, Ireland
Locations (8):
- Buenos Aires, Argentina
- Brazil (2):
  - Rio de Janeiro
  - São Paulo
- Chennai, India
- Kilifi, Kenya
- South Africa (3):
  - Durban
  - Johannesburg
  - Johannesburg Gauteng

REFERENCES:
- [Derived] Violari A, Bologna R, Kumarasamy N, Pilotto JH, Hendrickx A, Kakuda TN, Lathouwers E, Opsomer M, Van de Casteele T, Tomaka FL. Safety and efficacy of darunavir/ritonavir in treatment-experienced pediatric patients: week 48 results of the ARIEL trial. Pediatr Infect Dis J. 2015 May;34(5):e132-7. doi: 10.1097/INF.0000000000000644. PMID 25719453

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 5 countries: Argentina, Brazil, India, Kenya, and South Africa.
Pre-assignment Details: 27 participants were recruited and treated in this study; as Good Clinical Practice (GCP) requirements were not consistently adhered to at one site (involving 6 participants), analyses were performed excluding the participants from this site, resulting in 21 participants used for analyses.
Groups:
- DRV/Rtv: Before dose adjustment, oral darunavir suspension (100 mg/mL): 20 mg per kg body weight twice daily for children weighing between 10 and <20 kg. After dose adjustment, 25 mg per kg body weight twice daily if weight less than 15 kg, and fixed dose of 375 mg twice daily if weight more than or equal to 15 kg. Before dose adjustment, oral ritonavir solution (80 mg/mL): 3 mg per kg body weight twice daily and after dose adjustment fixed dose of 50 mg twice daily if weight more than or equal to 15 kg
Period: Overall Study
Arm/Group | DRV/Rtv
Started | 21
Completed | 20 ('Completed' represents the patients that are ongoing at the time of cut-off for the Week 24 analysis)
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | DRV/Rtv
Number analyzed (Participants) | 21
Age, Continuous [Median (Full Range); unit: years] | 4.6 (0.89) [3.2 to 5.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 10
Region of Enrollment [Number; unit: participants]
  Argentina | 4
  Brazil | 6
  India | 1
  South Africa | 10
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 15.1 (1.51)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Virological Response (Viral Load Less Than 50 Copies/mL) at Week 24 - Time to Loss of Virologic Response (TLOVR)
Description: The TLOVR algorithm was used to derive response, ie, response and loss of response needed to be confirmed at 2 consecutive visits and participants who permanently discontinued were considered nonresponders after discontinuation. Participants with intermittent missing viral load values were considered responders if the preceeding and succeeding visits indicated response. In all other cases, intermittent values were imputed with nonresponse. Resuppression after confirmed virologic failure was considered as failure in this algorithm.
Time Frame: Week 24
Population: 27 participants were recruited and received at least 1 dose of study medication; as Good Clinical Practice (GCP) requirements were not consistently adhered to at one site (involving 6 participant), analyses were performed excluding the participants from this site, resulting in 21 participants used for analyses.
Measure: Number; unit: Participants
Arm/Group | DRV/Rtv
Number analyzed (Participants) | 21
Participants | 13

2. Secondary Outcome: Number of Participants With Virological Response (Viral Load Less Than 50 Copies/mL) at Week 48
Time Frame: Week 48
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | DRV/Rtv
Number analyzed (Participants) | 21
Participants | 17

3. Secondary Outcome: Number of Participants With Virological Response (Viral Load Less Than 400 Copies/mL) at Week 24 and Week 48
Time Frame: Week 24 and Week 48
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | DRV/Rtv
Number analyzed (Participants) | 21
Participants
  Week 24 | 17
  Week 48 | 18

4. Secondary Outcome: Number of Participants With Less Than or Equal to 1 log10 Decrease in Plasma Viral Load at Week 24 and Week 48
Time Frame: Week 24 and Week 48
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | DRV/Rtv
Number analyzed (Participants) | 21
Participants
  Week 24 | 17
  Week 48 | 19

5. Secondary Outcome: Mean Change From Baseline to Week 24 and Week 48 in Plasma log10 Viral Load
Time Frame: Baseline, Week 24 and Week 48
Population: as for outcome 1
Measure: Mean (Standard Error); unit: log10 copies/mL
Arm/Group | DRV/Rtv
Number analyzed (Participants) | 21
log10 copies/mL
  Week 24 | -2.04 (0.244)
  Week 48 | -2.14 (0.257)

6. Secondary Outcome: Mean Change From Baseline to Week 24 and Week 48 in CD4+ Percentage
Time Frame: Baseline, Week 24 and Week 48
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Percentage of lymphocytes
Arm/Group | DRV/Rtv
Number analyzed (Participants) | 21
Percentage of lymphocytes
  Week 24 | 4 (0.9)
  Week 48 | 4 (1.3)

ADVERSE EVENTS:
Time Frame: 48 weeks
Arm/Group | DRV/Rtv
Serious Adverse Events (participants affected / at risk) | 2/21
Other Adverse Events (participants affected / at risk) | 18/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DRV/Rtv (N=21)
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 1
Trigger finger (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DRV/Rtv (N=21)
Neutropenia (Blood and lymphatic system disorders) | 2
Otitis media acute (Infections and infestations) | 2
Pharyngitis (Infections and infestations) | 2
Pyrexia (General disorders) | 3
Tachycardia (Cardiac disorders) | 2
Upper respiratory tract infection (Infections and infestations) | 6
Tinea capitis (Infections and infestations) | 5
Nasopharyngitis (Infections and infestations) | 4
Impetigo (Infections and infestations) | 3
Rhinitis (Infections and infestations) | 3
Lower respiratory tract infection (Infections and infestations) | 2
Otitis media chronic (Infections and infestations) | 2
Tinea faciei (Infections and infestations) | 2
Tonsillitis (Infections and infestations) | 2
Varicella (Infections and infestations) | 2
Diarrhoea (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 4
Dental caries (Gastrointestinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 3
Ear pain (Ear and labyrinth disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days